CLINICAL TRIAL: NCT03506438
Title: Addressing Palliative Care Needs Among Intensive Care Unit Family Members
Acronym: ICUconnect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00090202; 1U54MD012530 (NIH)
Record Dates: First submitted 2018-04-09; First posted 2018-04-24 (Actual); Results first posted 2023-11-13 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-10

CONDITIONS: Critical Illness; Family Members; Psychological Distress; Informal Caregivers; Palliative Care
Keywords: critical illness; palliative care; mobile app; psychological distress; depression; anxiety; informal caregiver
MeSH Terms: conditions — Critical Illness; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Unit of randomization is the ICU attending physician. We anticipate 15-25 ICU physicians for intervention and 15-25 for control. Therefore each clinician will likely have 5-12 family members each.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The electronic study data system login/password arrangement will not allow any investigator to ascertain treatment group.
  The study data system will automatically send links to study surveys for participant self-completion, and therefore outcomes assessors will be blinded to the majority of post-randomization data collection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ICU physician mobile app group (Experimental): Clinicians and family members will receive access to versions of the needs-focused mobile app that differ in content.
  Interventions: Behavioral: Needs-focused mobile app
- ICU physician usual care group (Placebo Comparator): Usual ICU care in an ICU as per the standards of the ICU attending
  Interventions: Other: Usual care

INTERVENTIONS:
Behavioral: Needs-focused mobile app — A mobile web app designed to assist both ICU clinicians in addressing patient/family needs and families in reporting their unmet needs.
  Arms: ICU physician mobile app group
Other: Usual care — Usual ICU care as per the standards of the ICU attending
  Arms: ICU physician usual care group

SUMMARY:
The quality of palliative care is highly variable for many patients treated in intensive care units (ICUs) and their family members. To address these challenges, the investigators will test the impact of a mobile app designed to help families navigate ICU-based palliative care vs. usual care. The investigators hypothesize that the intervention will reduce patient/family member unmet palliative care needs and improve the quality of clinical-family communication in racially/ethnically diverse populations.

DETAILED DESCRIPTION:
The quality of palliative care is highly variable in an intensive care unit (ICU) setting. These markers of poor quality are even more common among Black patients and families than among Whites. To address these challenges, the investigators developed a mobile app that allows families to both give and receive information relevant to palliative care and for ICU clinicians to visualize patient/family data and therefore better support them.

To determine the effect of this intervention,the investigators propose to conduct a randomized clinical trial (RCT) comparing the intervention to usual care to address four specific aims: (1) Using a cluster randomized clinical trial, determine the effect of the intervention vs usual care on unmet needs, psychological distress symptoms, and patient-centered care; (2) Determine the impact of the intervention on unmet needs and patient-centered care based across different racial groups; and (3) Explore family member and clinician experiences with intervention using mixed methods to understand mechanisms within unique case contexts [exploratory aim]. The investigators hypothesize that compared to usual care, ICUconnect will reduce family members' unmet needs, reduce family member psychological distress, increase the patient-centeredness care, and reduce hospital length of stay overall--though the magnitude of effect will be greater among Blacks compared to Whites

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* ≥18 years of age
* Receive mechanical ventilation in a study ICU for ≥48 hours under care of a study ICU physician

Exclusion Criteria (pre-consent):

* Decisional capacity
* Death expected within 24 hours
* Admission to an ICU at the index hospital >14 days
* Comfort care or withdrawal of treatment planned
* Imprisoned
* Extubated and possess decisional capacity prior to informed consent
* Died before T2 survey complete
* No known family or surrogate
* Care assumed by a non-study ICU attending after consent by patient/family but before T1
* Care assumed by non-study ICU attending <3 days after T1 but before T2
* Study ICU attending physicians from different groups (i.e., intervention or control) caring for patient change <3 days after T1 completed by family

Exclusion Criteria (post-consent):

* Patient regains decision making capacity before T2
* Patient dies before T2

FAMILY MEMBER

Inclusion Criteria:

* ≥18 years of age
* Self-described as the individual (related or unrelated) who provides the most support and with whom the patient has a significant relationship (per definition of 'family' described in the Society of Critical Care Medicine 2016 Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU)

Exclusion Criteria (pre-consent):

* Lack a knowledge of English such that the potential participant is not confident that they could complete study tasks (app viewing, surveys)
* Imprisoned
* Unable to complete surveys for any reason
* Describe their race as neither White nor Black*
* Describe their ethnicity as Hispanic*

  * Note that this study explicitly targets issues of racial disparities in healthcare, particularly of Black / African-Americans. Hispanics are excluded because of the pervasive nature of US residents' general belief that 'Hispanic' is a racial category.

Exclusion criteria (post-consent):

* If the assigned randomized ICU attending physician either leaves ICU service or is replaced by a non-participating ICU physician <= 2 calendar days after family member completes T1 survey
* Low need burden (NEST score <15)*

ICU PHYSICIANS

Inclusion Criteria:

* ≥18 years of age
* Attending physician in a study ICU

Exclusion Criteria:

- None

*The NEST score cutoff was changed on June 26, 2019. At this point, 3 patients had been randomized. This change was based on our review of data (NEST + psychological distress symptoms) from a parallel cohort study of >50 family members of ICU patients who met nearly identical eligibility criteria as for the ICUconnect trial. This was a larger cohort than the pilot study on which we based the NEST cutoff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-05-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cox, MD', Principal Investigator — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cox CE, Ashana DC, Riley IL, Olsen MK, Casarett D, Haines KL, O'Keefe YA, Al-Hegelan M, Harrison RW, Naglee C, Katz JN, Yang H, Pratt EH, Gu J, Dempsey K, Docherty SL, Johnson KS. Mobile Application-Based Communication Facilitation Platform for Family Members of Critically Ill Patients: A Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2349666. doi: 10.1001/jamanetworkopen.2023.49666. PMID 38175648

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a cluster randomized trial with randomization at the level of the ICU physician. Cluster size was 4 family member-patient dyads (2 Black and 2 White family members). Patients were used to determine family member eligibility.
Pre-assignment Details: Family members were excluded post-enrollment if their baseline NEST score was <15, representing low needs.
Groups:
- Family Members in ICU Attending Physician Mobile App Group; Patients in ICU Attending Mobile App Group; ICU Attendings in the ICU Attending Mobile App Group: Clinicians and family members will receive access to versions of the needs-focused mobile app that differ in content.
  Needs-focused mobile app: A mobile web app designed to assist both ICU clinicians in addressing patient/family needs and families in reporting their unmet needs.
- Family Members in ICU Attending Physician Usual Care Group; Patients in the ICU Attending Usual Care Group; ICU Attendings in the ICU Attending Usual Care Group: Usual ICU care
  Usual care: Usual ICU care is usual care from an ICU attending physician in an ICU setting, as per normal
Period: Overall Study
Arm/Group | Family Members in ICU Attending Physician Mobile App Group | Family Members in ICU Attending Physician Usual Care Group | Patients in ICU Attending Mobile App Group | Patients in the ICU Attending Usual Care Group | ICU Attendings in the ICU Attending Mobile App Group | ICU Attendings in the ICU Attending Usual Care Group
Started | 55 | 56 | 55 | 56 | 19 | 18
Completed | 47 | 49 | 47 | 49 | 19 | 18
Not Completed | 8 | 7 | 8 | 7 | 0 | 0
Not completed — Lost to Follow-up | 8 | 7 | 8 | 7 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Family members of patients managed in an ICU, patients managed in an ICU, and ICU attending physicians working in adult ICUs.
Groups:
- Family Members in ICU Attending Physician Usual Care Group; Patients in ICU Attending Usual Care Group; ICU Attendings in the ICU Attending Usual Care Group: Usual ICU care
  Usual care: Usual ICU care is standard care from an ICU attending in an ICU setting per the standards of the care area without a mobile app
- Patients in ICU Attending Physician Mobile App Group; ICU Attendings in the ICU Attending Mobile App Group: Clinicians and family members will receive access to versions of the needs-focused mobile app that differ in content.
  Needs-focused mobile app: A mobile web app designed to assist both ICU clinicians in addressing patient/family needs and families in reporting their unmet needs.
- Total: Total of all reporting groups
Arm/Group | Family Members in ICU Attending Physician Mobile App Group | Family Members in ICU Attending Physician Usual Care Group | Patients in ICU Attending Physician Mobile App Group | Patients in ICU Attending Usual Care Group | ICU Attendings in the ICU Attending Mobile App Group | ICU Attendings in the ICU Attending Usual Care Group | Total
Number analyzed (Participants) | 55 | 56 | 55 | 56 | 19 | 18 | 259
Age, Continuous [Median (Inter-Quartile Range); unit: years] — Population: Age was not collected for ICU attending physicians.
  years
    number analyzed (Participants) | 55 | 56 | 55 | 56 | 0 | 0 | 222
    (all) | 51 [43 to 58] | 54 [43 to 62] | 55.7 [44 to 62.9] | 57.9 [46 to 67.6] |  |  | 54.7 [44 to 62.6]
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Gender self-described as man | 12 | 7 | 28 | 38 | 12 | 11 | 108
  Gender self-described as woman | 43 | 49 | 27 | 18 | 7 | 7 | 151
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — This trial only enrolled non-Hispanic White and Black family members given the focus on racial disparities.
  Participants
    Hispanic or Latino | 0 | 0 | 0 | 0 | 1 | 2 | 3
    Not Hispanic or Latino | 55 | 56 | 55 | 56 | 18 | 16 | 256
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 19 | 28 | 18 | 27 | 0 | 0 | 92
  White | 36 | 28 | 36 | 29 | 15 | 16 | 160
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 55 | 56 | 55 | 56 | 19 | 18 | 259
Needs; existential concerns; symptoms; and therapeutic interaction (NEST) scale [Mean (Standard Deviation); unit: units on a scale] — This is a measure completed by family members (not patients and not ICU physicians) that assesses palliative care need across 8 domains of palliative care quality. It is the primary study outcome. Population: Note that the NEST was completed by family members only in this study (i.e., NOT by patients and NOT by ICU physicians). For this reason, these sections are blank.
  units on a scale
    number analyzed (Participants) | 55 | 56 | 0 | 0 | 0 | 0 | 111
    (all) | 36.9 (19.0) | 36.3 (17.4) |  |  |  |  | 37.0 (18.0)

OUTCOME MEASURES:

1. Primary Outcome: Needs; Existential Concerns; Symptoms; and Therapeutic Interaction (NEST) Scale Total Score
Description: A palliative care needs instrument that assesses palliative care needs across all 8 domains of palliative care quality. Scores on this 13-item instrument can range from 0 (no needs) to 130 (higher needs)
Time Frame: Time 1 (baseline), Time 2 (target ~3 days post-randomization), and Time 3 (target ~1 week post-randomization)
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Family Members in the ICU Attending Mobile App Group: Clinicians and family members will receive access to versions of the needs-focused mobile app that differ in content.
  Needs-focused mobile app: A mobile web app designed to assist both ICU clinicians in addressing patient/family needs and families in reporting their unmet needs.
- Family Members in the ICU Attending Usual Care Group: Usual ICU care
  Usual care: Usual ICU care per the standards of the ICU attending
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
score on a scale
  NEST baseline | 36.9 (19.0) | 36.3 (17.4)
  NEST day 3 | 26.5 (19.1) | 32.3 (22.1)
  NEST day 7 | 24.9 (19.5) | 29.6 (20.2)
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.018, Mixed Models Analysis; Mean Difference (Net) = -6.7, 95% CI 2-sided [-12.2 to -1.2]

2. Secondary Outcome: Patient Health Questionnaire 9-Item Scale (PHQ-9)
Description: A depression symptoms instrument. Scores range from 0 (no depression symptoms) to 27 (higher depression symptoms)
Time Frame: Time 1 (baseline), Time 2 (target ~3 days post-randomization), and Time 4 (3 months post-randomization)
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
score on a scale
  PHQ-9 baseline | 8.0 (3.5) | 7.7 (3.6)
  PHQ-9 day 3 | 6.9 (3.7) | 6.4 (3.1)
  PHQ-9 3 months | 6.0 (3.4) | 6.0 (3.4)
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Net) = 0.3, 95% CI 2-sided [-0.5 to 1.1]

3. Secondary Outcome: Generalized Anxiety Disorder 7-Item Scale (GAD-7)
Description: An anxiety symptoms instrument. Scores range from 0 (no anxiety symptoms) to 21 (higher anxiety symptoms)
Time Frame: Time 1 (baseline), Time 2 (target ~3 days post-randomization), and Time 4 (3 months post-randomization)
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Family Members in the ICU Attending Usual Care Group: Usual ICU care
  Usual care: Usual ICU care per the standard of the ICU attending
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
score on a scale
  GAD-7 baseline | 9.2 (6.3) | 8.4 (5.9)
  GAD-7 3 days | 7.9 (6.1) | 7.4 (5.4)
  GAD-7 month 3 | 6.1 (5.2) | 5.3 (5.0)
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.73, Mixed Models Analysis; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-1.4 to 1.0]

4. Secondary Outcome: Post-Traumatic Stress Symptom (PTSS) Inventory
Description: A post-traumatic stress disorder symptom instrument. Scores range from 10 (low PTSD symptoms) to 70 (higher PTSD symptoms)
Time Frame: Time 1 (baseline) and Time 4 (3 months post-randomization)
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
score on a scale
  PTSS baseline | 26.2 (14.8) | 24.5 (13.6)
  PTSS month 3 | 25.4 (15.7) | 23.0 (13.9)
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.47, Mixed Models Analysis; estimated mean difference = 0.6, 95% CI 2-sided [-1.0 to 2.1]

5. Secondary Outcome: Number of Participants With Goal Concordant Care
Description: A measure of the alignment between patient values and treatments received. This is a dichotomous scale; care is either concordant or discordant.
Time Frame: Time 1 (baseline) and Time 2 (target ~3 days post-randomization)
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
Participants
  Baseline | 37 | 50
  Day 3 | 47 | 47
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.29, Regression, Logistic; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.6 to 5.2]

6. Secondary Outcome: Post-randomization Hospital Length of Stay (Days)
Description: Patient hospital length of stay measured in days post-randomization
Time Frame: Across the entire hospitalization after randomization (approximately 2 months)
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
days | 37.2 (21.2) | 38.6 (21.2)
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.47, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Post-randomization Intensive Care Unit Length of Stay (Days)
Description: Patient intensive care unit length of stay post-randomization
Time Frame: Across the entire hospitalization after randomization (approximately 2 months)
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
days | 21.2 (16.4) | 21.2 (12.0)
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.39, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Participants Who Responded "Usually" or "Always" on the Interpersonal Processes of Care 18-Item (IPC-18) Short Form Scale - Communication Domain
Description: The IPC-18 is a measure of the interpersonal aspects of care. Interpersonal processes of care are the social-psychological aspects of the patient-physician interaction. These components of quality of care may help explain disparities in health between minority patients and their counterparts. The "elicited concerns, responded" scale within the Communication domain is used here. All items use an identical set of response options: 1='never'; 2='rarely'; 3='sometimes'; 4='usually'; 5='always.' A higher score indicates better processes.
Time Frame: Baseline (at time of randomization) and ~3 days post-randomization
Population: Data not collected on the the patient and ICU attendings Arms/Groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Family Members in the ICU Attending Mobile App Group | Family Members in the ICU Attending Usual Care Group
Number analyzed (Participants) | 55 | 56
Participants
  Day 1 | 46 | 47
  Day 3 | 49 | 44
Statistical Analysis 1: Comparison: Family Members in the ICU Attending Mobile App Group vs Family Members in the ICU Attending Usual Care Group; Test type: Superiority; p = 0.08, Regression, Logistic

ADVERSE EVENTS:
Time Frame: 3 months
Description: Note that adverse event data (death, hospitalization) was collected on patients included in the trial. Note also that patients were not formally included in the trial in the sense that they completed no surveys, etc., but rather were the starting point for ascertaining eligibility for their family members.
Groups:
- Patients in ICU Attending Physician Usual Care Group; Family Members in ICU Attending Physician Usual Care Group; ICU Attending in the ICU Attending Usual Care Group: Usual ICU care
  Usual care: Usual ICU care per the standards of the ICU attending
- ICU Attending in the ICU Attending Group: Clinicians and family members will receive access to versions of the needs-focused mobile app that differ in content.
  Needs-focused mobile app: A mobile web app designed to assist both ICU clinicians in addressing patient/family needs and families in reporting their
Arm/Group | Patients in ICU Attending Physician Mobile App Group | Patients in ICU Attending Physician Usual Care Group | Family Members in ICU Attending Physician Mobile App Group | Family Members in ICU Attending Physician Usual Care Group | ICU Attending in the ICU Attending Group | ICU Attending in the ICU Attending Usual Care Group
All-Cause Mortality (participants affected / at risk) | 17/55 | 15/56 | 0/55 | 0/56 | 0/19 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 0/55 | 0/56 | 0/19 | 0/18
Other Adverse Events (participants affected / at risk) | 0/55 | 0/56 | 0/55 | 0/56 | 0/19 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03506438/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-28): https://cdn.clinicaltrials.gov/large-docs/38/NCT03506438/SAP_001.pdf
  • Informed Consent Form (2022-01-20): https://cdn.clinicaltrials.gov/large-docs/38/NCT03506438/ICF_002.pdf